CLINICAL TRIAL: NCT04328012
Title: Comparison Of Therapeutics for Hospitalized Patients Infected With SARS-CoV-2 In a Pragmatic aDaptive randoMizED Clinical Trial During the COVID-19 Pandemic (COVID MED Trial)
Brief Title: COVID MED Trial - Comparison Of Therapeutics for Hospitalized Patients Infected With COVID-19
Acronym: COVIDMED
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: difficult enrollment
Sponsor: Bassett Healthcare (Other)
Collaborators: Reid Health (Unknown); Goshen Health System (Other)
Responsible Party: Principal Investigator, Daniel Freilich, MD, attending physician - hospitalist, Bassett Healthcare
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1581969
Record Dates: First submitted 2020-03-27; First posted 2020-03-31 (Actual); Last update posted 2022-03-24 (Actual); Status verified 2022-03

CONDITIONS: SARS-CoV-2 Infection
Keywords: COVID; COVID-19; coronavirus
MeSH Terms: conditions — COVID-19; Coronavirus Infections | interventions — Losartan

STUDY DESIGN:
Intervention Model Description: randomized, double blind, placebo controlled clinical trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Losartan (Experimental): losartan 25 mg po QD X 14 days
  Interventions: Drug: Losartan
- Placebo (Placebo Comparator): placebo QD X 14 days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Losartan — administered 14 days
  Other Names: Cozaar
  Arms: Losartan
Drug: Placebo — administered 14 days
  Arms: Placebo

SUMMARY:
In a randomized, double-blind, placebo-controlled, multi-center, Phase 2-like, investigator-directed trial, hospitalized adult patients with laboratory confirmed SARS-CoV-2 infection meeting inclusion and exclusion criteria, will be provided information on the trial, offered enrollment, and if informed consent provided, enrolled randomly in a 2:1 ratio to one of two groups: Group 1 standard care and losartan or Group 2 standard care and placebo. Patients will be followed for up to 60 days, with data collected to quantify the NCOSS over time (the primary objective), and for the trial's secondary objectives (see outcome measurements below).

DETAILED DESCRIPTION:
Although a number of therapeutics have been utilized by clinicians to treat hospitalized patients with COVID-19, none were systematically evaluated in clinical trials at the time of the outset of this RCT (COVID MED). Since then, dexamethasone has been shown to decrease mortality and remdesivir to possibly decrease hospital LOS in the RECOVERY and ACTT-II trials and others. The initial iteration of this protocol included 4 arms, hydroxychloroquine, lopinavir/ritonavir, losartan, and placebo based on suggestive efficacy and safety and widespread empiric use. The current iteration of COVID MED includes two arms, standard of care and losartan vs. standard of care and placebo.

Hydroxychloroquine was initially included in COVID MED based on suggestive in vitro, animal preclinical, and early RCT data, and widespread empiric use in hospitalized patients with COVID-19. Lopinavir/ritonavir, an antiretroviral medication, showed equivocal and possibly positive efficacy and safety in an early pandemic Chinese RCT published in NEJM. After public release and eventual publication of the negative results for hydroxychloroquine and then lopinavir/ritonavir initially from the RECOVERY trial and then others, enrollment in COVID MED in these two arms was halted and then discontinued permanently. Data from subjects enrolled in the hydroxychloroquine arm are being incorporated into a pooled analysis of RCTs by the Trial Innovation Network.

Losartan, an angiotensin II receptor blocker (ARB), has theoretical benefit as SARSCoV-2 appears to bind to lung tissue via Angiotensin-Converting Enzyme 2 (ACE-2) receptors which might be inhibited by ARBs; other potential benefits have been hypothesized as well. Since the initial iteration of this protocol, observational studies have shown that patients already taking ACEi/ARB medications do not have adverse outcome when these drugs are continued in hospitalized COVID-19 patients. These data have reinforced continuation of the losartan vs. placebo arms of this RCT which are ongoing.

This pragmatic adaptive trial continues to compare outcome in hospitalized COVID-19 patients treated with standard of care and losartan vs. standard of care and placebo.

ELIGIBILITY:
Inclusion criteria

1. Hospitalized patient
2. Age >= 18 years
3. Able to ingest oral medication or be administered medication via gastric tube or equivalent
4. Laboratory confirmation of SARS-CoV-2 infection within 1 week prior to randomization
5. Randomization within 72 hr of hospital admission
6. Negative pregnancy test for reproductive age women
7. Patient or LAR able to provide informed consent

Exclusion criteria

1. Allergy or intolerance to losartan or other ARBs
2. Already taking ACE or ARB (within 1 month)
3. Hypotension at time of enrollment (SBP < 100 mm Hg)
4. Hyperkalemia (K >/= 5.0 at time of screening or history of hyperkalemia)
5. Severe renal dysfunction (estimated GFR < 30 ml/min at time of screening or history advanced renal disease)
6. Severe volume depletion or acute kidney injury (AKI) at time of enrollment
7. Known cirrhotic ascites
8. Known severe aortic or mitral valve stenosis
9. Known unstented renal artery stenosis
10. Co-administration with certain drugs due to CYP3A interactions if taken in < 24 hr
11. Severe hepatic insufficiency (LFTs > 5 times the upper limit of normal or known ESLD or cirrhosis)
12. Nausea/vomiting or aspiration risk precluding oral medications unless can be given by gastric tube
13. Pregnancy or breast feeding
14. Absence of dependable contraception in reproductive age women
15. Inability to obtain or declined informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2020-04-06 (Actual); Primary Completion 2021-07-01 (Actual); Study Completion 2021-12-01 (Actual)

PRIMARY OUTCOMES:
National Institute of Allergy and Infectious Diseases COVID-19 Ordinal Severity Scale (NCOSS) | 60 days
  difference in NCOSS scores between the different treatment groups

SECONDARY OUTCOMES:
Hospital length of stay (LOS) | 60 days
  difference in the total inpatient LOS between the three treatment groups
Intensive care unit level LOS | 60 days
  difference in the total ICU level care LOS between the three treatment groups
Mechanical ventilation | 60 days
  difference in length of use of mechanical ventilation between the three treatment groups
survival | 60 days
  difference in all cause mortality between the four treatment groups

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Freilich, MD, Principal Investigator — Bassett Medical Center
Locations (1):
- Bassett Medical Center, Cooperstown, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kreuzberger N, Hirsch C, Chai KL, Tomlinson E, Khosravi Z, Popp M, Neidhardt M, Piechotta V, Salomon S, Valk SJ, Monsef I, Schmaderer C, Wood EM, So-Osman C, Roberts DJ, McQuilten Z, Estcourt LJ, Skoetz N. SARS-CoV-2-neutralising monoclonal antibodies for treatment of COVID-19. Cochrane Database Syst Rev. 2021 Sep 2;9(9):CD013825. doi: 10.1002/14651858.CD013825.pub2. PMID 34473343